CLINICAL TRIAL: NCT00767611
Title: Molecular Markers of Human Sperm Function
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909001; 09-E-N001
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Infertility; Reproduction; Reproductive Techniques, Assisted
Keywords: Infertility; Sperm; Embryo Development; In Vitro Fertilization
MeSH Terms: conditions — Infertility; Helping Behavior

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objectives:

Male factor infertility is poorly understood and our ability to evaluate the male contribution to a couple's infertility is very limited. The overarching goal of this project is to understand at the molecular level what functional activities in human sperm are required for successful fertilization leading to full term development. These findings will allow us to develop new methods to determine the impact of environmental exposures on sperm quality and male fertility.

A sperm protein known as phospholipase C zeta (PLC zeta) initiates embryo development at fertilization. The primary objective of this study is to test the hypothesis that human PLC zeta activity correlates directly with the proportion of fertilized eggs that undergo early cleavage during an in vitro fertilization (IVF) cycle. Secondary objectives for the study are to generate preliminary data regarding the variability in sperm PLC zeta activity within and between individuals and to determine if there are clinical or laboratory correlates for sperm PLC zeta activity.

Study population:

The study population will consist of 178 infertile couples undergoing IVF procedures at Duke Fertility Center (DFC) from which we will obtain 154 evaluable couples for the study.

Overall Design:

An observational cohort study design will be used to assess the association of PLC zeta activity in the residual sperm from the sample used for an IVF cycle with the proportion of eggs per couple that undergo early cleavage during the same cycle. Infertile couples enrolling in an IVF treatment cycle at DFC will be approached for inclusion in the study. Consent will be obtained from both male and female partners, and historical medical information and information about their IVF cycle will be collected by chart review. Blood for isolation of serum and DNA will be collected only from the male partner for evaluation of hormone levels and genetic analyses related to infertility. On the day of the egg retrieval, residual sperm not needed for clinical purposes will be transported via courier to NIEHS. Sperm PLC zeta activity will be measured in the investigator's laboratory using an experimental bioassay. Sperm PLC zeta protein will be analyzed at the University of Massachusetts.

Outcome Parameters:

The primary outcome will be the proportion of embryos that undergo early cleavage. Secondary outcomes will include proportion of eggs fertilized, embryo development parameters, and p...

DETAILED DESCRIPTION:
Objectives:

Male factor infertility is poorly understood and our ability to evaluate the male contribution to a couple's infertility is very limited. The overarching goal of this project is to understand at the molecular level what functional activities in human sperm are required for successful fertilization leading to full term development. These findings will allow us to develop new methods to determine the impact of environmental exposures on sperm quality and male fertility.

A sperm protein known as phospholipase C zeta (PLC zeta) initiates embryo development at fertilization. The primary objective of this study is to test the hypothesis that human PLC zeta activity correlates directly with the proportion of fertilized eggs that undergo early cleavage during an in vitro fertilization (IVF) cycle. Secondary objectives for the study are to generate preliminary data regarding the variability in sperm PLC zeta activity within and between individuals and to determine if there are clinical or laboratory correlates for sperm PLC zeta activity.

Study population:

The study population will consist of 178 infertile couples undergoing IVF procedures at Duke Fertility Center (DFC) from which we will obtain 154 evaluable couples for the study.

Overall Design:

An observational cohort study design will be used to assess the association of PLC zeta activity in the residual sperm from the sample used for an IVF cycle with the proportion of eggs per couple that undergo early cleavage during the same cycle. Infertile couples enrolling in an IVF treatment cycle at DFC will be approached for inclusion in the study. Consent will be obtained from both male and female partners, and historical medical information and information about their IVF cycle will be collected by chart review. Blood for isolation of serum and DNA will be collected only from the male partner for evaluation of hormone levels and genetic analyses related to infertility. On the day of the egg retrieval, residual sperm not needed for clinical purposes will be transported via courier to NIEHS. Sperm PLC zeta activity will be measured in the investigator's laboratory using an experimental bioassay. Sperm PLC zeta protein will be analyzed at the University of Massachusetts.

Outcome Parameters:

The primary outcome will be the proportion of embryos that undergo early cleavage. Secondary outcomes will include proportion of eggs fertilized, embryo development parameters, and pregnancy outcome. Association of PLC zeta activity with male partner's clinical or laboratory information will be determined. Variability in sperm PLC zeta activity will be determined within and between individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Infertile couples undergoing an ART cycle at DFC in which eggs are retrieved from the female partner. This type of ART cycle comprises approximately 80-90 percent of the ART cycles at DFC.
* Infertile couples undergoing an ART cycle at DFC in which the eggs are retrieved from an anonymous egg donor. Approximately 10-20 percent of the ART cycles at DFC involve anonymous egg donation.
* Willing and able to provide informed consent.
* Age greater than or equal to 18 (both partners in couple). Essentially all infertile couples who enter clinical ART programs at least age 18.

EXCLUSION CRITERIA:

* Previous completed participation in the study. A complete data set will be obtained from either partner of a couple only once for this study.
* Cancellation of the ART cycle prior to egg retrieval, or no fertilizable eggs retrieved. In this case it would not be possible to determine our primary outcome.
* Age less than 18 (either partner in couple). Because they so rarely experience clinical infertility, we do not expect any couples under age 18 to enter the ART program, so we will not include these as subjects.
* Use of frozen sperm to inseminate eggs. The rationale for this exclusion is that the effect of cryopreservation reagents on PLC zeta activity is unknown, and very few of the ART cycles at DFC utilize donor sperm so we would not be able to control appropriately for this confounder.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Chandra A, Martinez GM, Mosher WD, Abma JC, Jones J. Fertility, family planning, and reproductive health of U.S. women: data from the 2002 National Survey of Family Growth. Vital Health Stat 23. 2005 Dec;(25):1-160. PMID 16532609
- [Background] Esfandiari N, Javed MH, Gotlieb L, Casper RF. Complete failed fertilization after intracytoplasmic sperm injection--analysis of 10 years' data. Int J Fertil Womens Med. 2005 Jul-Aug;50(4):187-92. PMID 16405104
- [Background] Kouchi Z, Fukami K, Shikano T, Oda S, Nakamura Y, Takenawa T, Miyazaki S. Recombinant phospholipase Czeta has high Ca2+ sensitivity and induces Ca2+ oscillations in mouse eggs. J Biol Chem. 2004 Mar 12;279(11):10408-12. doi: 10.1074/jbc.M313801200. Epub 2003 Dec 29. PMID 14701816